CLINICAL TRIAL: NCT06902727
Title: Effects of Virtual Reality Exercise on Promoting Physical Activity and Health Among College Students: A 4-week Randomized Controlled Trial
Brief Title: Effects of Virtual Reality Exercise on Promoting Physical Activity and Health Among College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Principal Investigator, Zan Gao, Professor and Department Head, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00010580
Record Dates: First submitted 2025-03-03; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Physical Activity Levels; Cardiovascular Fitness; Body Composition; Situational Motivation; Situational Interest; Mood States; Depressive Symptoms
Keywords: Exergaming; Physical Activity; Virtual Reality; Video games; VR games; Physical Activity Levels; Cardiovascular fitness
MeSH Terms: conditions — Depression; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise on immersive VR-based bike (Experimental): Participants were asked to exercise on an immersive VR-based exercise bike for one hour per session, two times per week, for 4 weeks
  Interventions: Device: VR-based exercise bike
- Usual routine (Active Comparator): Participants in the control group were asked to maintain their usual routine after the baseline test for 4 weeks. Participants were scheduled separately coming to lab for the post-test after 4 weeks and all participants received the identical assessments in aforementioned physiological and psychological outcomes.
  Interventions: Other: Usual routine

INTERVENTIONS:
Device: VR-based exercise bike — For the intervention group, participations exercised on an immersive VR-based exercise bike for one hour, twice per week, for 4 weeks. Participants in the control group were asked to maintain their usual routine after the baseline test for 4 weeks. Participants were scheduled separately coming to lab for the post-test after 4 weeks and all participants received the identical assessments in aforementioned physiological and psychological outcomes.
  Arms: Exercise on immersive VR-based bike
Other: Usual routine — Participants were asked to maintain their usual activities, without engaging in any other physical activity intervention during the 4-week study period.
  Arms: Usual routine

SUMMARY:
The purpose of this research is to examine the effectiveness of a 4-week immersive-virtual reality (VR) exercise bike intervention on college students' physiological outcomes (physical activity levels, cardiovascular fitness, and body composition) and psychological outcomes (situational motivation, situational interest, mood states, and depressive symptoms).

ELIGIBILITY:
Inclusion Criteria:

* College students age from 18 to 35 years old who are currently enrolled in the university
* College students without diagnosed physical and/or mental disabilities
* Must be willing to provide informed consent and compete the PA Readiness Questionnaire (PAR-Q)
* Must be willing to be randomized into an intervention or control group
* no self-reported motion sickness symptoms during immersive VR-based exercise

Exclusion Criteria:

* Students under the age of 18 or over the age of 35 years old or not currently enrolled in the university
* Having self-reported physical and/or mental disabilities
* Contradictions to PA participation as determined by PAR-Q responses
* having motion sickness reaction when exercising under VR-based condition.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Exercise Motivation | Baseline, and 4 weeks
  Participants' motivation were assessed by the Behavioral Regulation in Exercise Questionnire-2 (BREQ-2). The BREQ-2 has 19 items assessing the continuum of behavioral regulation in exercise, which included amotivation, external regulation, introjected regulation, identified regulation, and intrinsic regulation.
Mood States | Baseline, and 4 weeks
  Participants' mood states were measured by the Brunel Mood Scale (BRUMS). The BRUMS assesses mood across six subscales (anger, confusion, depression, fatigue, tension, and vigor) using a 24-item questionnaire with responses ranging from 0 (not at all) to 4 (extremely).
Depressive Symptoms | Baseline, and 4 weeks
  The Beck Depression Inventory (BDI) was used to assess participant's depressive symptoms. This is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. The total score was calculated to the evaluate the severity of depressive symptoms.

SECONDARY OUTCOMES:
Cardiovascular fitness levels | Baseline, and 4 weeks
  Investigators asked participants to step on and off of a 12-inch plyometric box for 3 minutes to the "beep" of a metronome set to 96 beats-per-minute, with each beep corresponding with one leg movement. Immediately following the completion of the test, the principal investigator measured participants' heart rate for 60 seconds via palpation of the radial artery on the underbelly of the left wrist.
Physical activity levels | Baseline, and 4 weeks
  Physical activity levels were assessed via International Physical Activity Questionnaire (IPAQ). The IPAQ assesses three specific types of activity: walking, moderate-intensity activities, and vigorous-intensity activities. It asks participants to recall the time (in minutes) spent on each of these activities in the past 7 days.
  Each participant were assigned an accelerometer to wear during each 60-minute exercise session. Prior to the start of the intervention, participants were asked to wear an accelerometer for one week for measuring their physical activity levels. In addition, the investigators asked participants to wear the accelerometer for another week at the completion of 4-week intervention.
Body Mass Index | Baseline, and 4 weeks
  Participant height (cm) and weight (kg) were measured using a stadiometer and a Tanita BC-558 IRONMAN Segmental Body Composition Monitor, respectively, in theUniversity of Minnesota's Physical Activity Epidemiology Laboratory. Both height and weight were used to calculate BMI in kg/m². BMI was classified according to the following indicators: Underweight: BMI < 18.5; Normal weight: BMI 18.5-24.9; Overweight: BMI 25-29.9; Obesity: BMI ≥ 30.
Percent of body fat | Baseline, and 4 weeks
  Percent of body fat (%BF) were measured by Tanita BC-558 IRONMAN Segmental Body Composition Monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Twin Cities, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data, including primary and secondary outcomes, and relevant demographic will be made publicly available. Data will be accessible through a public data repository. Researchers interested in accessing these datasets can request or directly download them via https://www.openicpsr.org/openicpsr/project/223741/version/V1/view

REFERENCES:
- [Derived] Liu W, McDonough DJ, Oginni J, Mavoungou J, Gao Z. Effects of an Immersive Virtual Reality-Based Exercise Intervention on Psychological and Physiological Outcomes in College Students: Randomized Controlled Trial. JMIR Serious Games. 2025 Dec 15;13:e75777. doi: 10.2196/75777. PMID 41307454